CLINICAL TRIAL: NCT04232215
Title: Feasibility and Acceptability of a Medical Grade, Smartphone-based, Fetal Heart Rate Monitor for Outpatient Use: the HeraBEAT™ Clinical Trial
Brief Title: Medical Grade, Smartphone-based, Fetal Heart Rate Monitor for Outpatient Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yvonne S. Butler Tobah, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-004708
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Intervention Model Description: After approximately 8 weeks of monitoring, patients will complete an ease of use survey, then crossover to the alternate study product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- HeraBEAT™ Intervention Group (Experimental): Subjects will monitor their fetal heart beat once weekly using the HeraBEAT™ device. After approximately 8 weeks of monitoring subjects will crossover to using the doppler fetal heart rate monitor
  Interventions: Device: HeraBEAT™
- Standard Fetal Doppler Group (Active Comparator): Subjects will monitor their fetal heart beat once weekly using the doppler fetal heart rate monitor. After approximately 8 weeks of monitoring subjects will crossover to using the HeraBEAT™ device
  Interventions: Device: Doppler fetal heart rate monitor

INTERVENTIONS:
Device: HeraBEAT™ — A wireless Smart Fetal Ultrasound Doppler measuring device designed to be self-administered by the expectant mother throughout the different stages of pregnancy
  Arms: HeraBEAT™ Intervention Group
Device: Doppler fetal heart rate monitor — A hand-held ultrasound transducer that uses the Doppler Effect to provide an audible simulation of the heart beat and displays the number of beats per minute.
  Arms: Standard Fetal Doppler Group

SUMMARY:
Researchers are assessing the ease of use and accuracy of the HeraBEAT™ device, a new device used with a smartphone to monitor fetal heart rate during pregnancy.

DETAILED DESCRIPTION:
The HeraBEAT™ is a wireless Smart Fetal Ultrasound Doppler measuring device designed to be self-administered by the expectant mother throughout the different stages of pregnancy. The HeraBEAT™ device safety and performance claims allow continuous and accurate measurement of fetal heart rate (FHR) and maternal heart rate (MHR) throughout the pregnancy starting at 12 weeks gestation.

Technologically, HeraBEAT™ is similar to other FHR devices currently on the market in terms of device usage but differ by design in its interface. The HeraBEAT™ device uses a smartphone-based interface, with real time instructions for expectant mothers for determining both MHR and FHR.

This study will recruit low risk expectant mothers from the Obstetrics and Gynecology Department at Mayo Clinic Rochester. This is a mixed method; single center randomized controlled trial comparing HeraBEAT™ to a standard home fetal Doppler monitor, in the outpatient setting at a single academic institution, in the mid-west United States. The overall study will be guided by an assessment of device functionality and user acceptability, as well as an evaluation of the impact of the device on expectant mother's perception of fetal well-being, as measured by standardized surveys.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to speak, read and understand English
* Able to provide informed consent
* Owns a suitable iOS or Android device and demonstrates average control and basic understanding of using a smartphone
* At least 12 weeks gestation
* Pregnancy documented as low risk

Exclusion Criteria:

* Any observed anomalies on first trimester dating or formal ultrasound
* Multifetal gestation
* Maternal history of defibrillation
* Maternal history of electro-surgery
* Patients with external electrical stimulators, cardiac pacemakers or requiring use of MRI or other high frequency medical equipment
* Clinical judgment that determines that the pregnancy is at high risk for complications
* Any of the following high risk factors would disqualify the mother for the study:

  * Abnormal fetal anatomy
  * Chronic hypertension, including severe hypertension (>160/110)
  * Possible ectopic pregnancy or pregnancy of unknown location
  * Multi-fetal pregnancy
  * Hypertensive disorders (chronic hypertension, gestational diabetes, preeclampsia)
  * Prior Pulmonary Embolism / Deep Vein Thrombosis / stroke
  * Anticoagulation during prior pregnancy (e.g. antiphospholipid antibody syndrome)
  * Prosthetic heart valve (non-bio)
  * Pulmonary hypertension
  * Mothers currently taking Immunosuppressants, Prednisone > 10mg per day)
  * Women with mental health disorders (including eating disorders, severe depression, on antipsychotics)
  * Recurrent pregnancy loss (>2 losses)
  * Current maternal malignancy
  * Prior myocardial infarction/cardiomyopathy
  * Bio-prosthetic heart valves
  * Marfan syndrome
  * Active liver disease (e.g. hepatitis)
  * Congenital heart disease
  * Coagulopathies including thrombophilias and bleeding disorders.
  * Pre-existing diabetes
  * Genetic disease/Cystic Fibrosis testing/anomalies in prior child
  * Incompetent cervix (prior cerclage)
  * Isoimmunization (Rh, Kell, etc.)
  * History of transplant or currently on Dialysis
  * Prior 2nd or 3rd trimester loss
  * Human Immunodeficiency Virus (HIV)
  * Inflammatory bowel disease
  * Asthma and currently on steroid to control disease
  * History of preterm delivery <37 weeks
  * BMI >40 (class 3 obesity)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne S Butler Tobah, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants will be asked to discontinue the study if their pregnancy is subsequently diagnosed as high risk, or if cardiac or cranial anomalies are identified on routine fetal sonography. 4 of the 59 patients enrolled (i.e. signed consent) were not randomized and therefore withdrawn from the study,
Groups:
- HeraBEAT™ Intervention Group, Then Standard Fetal Doppler: Subjects will monitor their fetal heart beat once weekly using the HeraBEAT™ device. After approximately 8 weeks of monitoring subjects will crossover to using the doppler fetal heart rate monitor
  HeraBEAT™: A wireless Smart Fetal Ultrasound Doppler measuring device designed to be self-administered by the expectant mother throughout the different stages of pregnancy
- Standard Fetal Doppler Group, Then HeraBEAT™ Intervention: Subjects will monitor their fetal heart beat once weekly using the doppler fetal heart rate monitor. After approximately 8 weeks of monitoring subjects will crossover to using the HeraBEAT™ device
  Doppler fetal heart rate monitor: A hand-held ultrasound transducer that uses the Doppler Effect to provide an audible simulation of the heart beat and displays the number of beats per minute.
Period: First Intervention (8 Weeks)
Arm/Group | HeraBEAT™ Intervention Group, Then Standard Fetal Doppler | Standard Fetal Doppler Group, Then HeraBEAT™ Intervention
Started | 28 | 27
Completed | 28 | 25
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention (8 Weeks)
Arm/Group | HeraBEAT™ Intervention Group, Then Standard Fetal Doppler | Standard Fetal Doppler Group, Then HeraBEAT™ Intervention
Started | 28 | 25
Completed | 28 | 1
Not Completed | 0 | 24

BASELINE CHARACTERISTICS:
Groups:
- HeraBEAT™ Intervention, Then Standard Fetal Doppler Group: Subjects will monitor their fetal heart beat once weekly using the HeraBEAT™ device. After approximately 8 weeks of monitoring subjects will crossover to using the doppler fetal heart rate monitor
  HeraBEAT™: A wireless Smart Fetal Ultrasound Doppler measuring device designed to be self-administered by the expectant mother throughout the different stages of pregnancy
- Standard Fetal Doppler Then HeraBEAT™ Intervention Group: Subjects will monitor their fetal heart beat once weekly using the doppler fetal heart rate monitor. After approximately 8 weeks of monitoring subjects will crossover to using the HeraBEAT™ device
  Doppler fetal heart rate monitor: A hand-held ultrasound transducer that uses the Doppler Effect to provide an audible simulation of the heart beat and displays the number of beats per minute.
- Total: Total of all reporting groups
Arm/Group | HeraBEAT™ Intervention, Then Standard Fetal Doppler Group | Standard Fetal Doppler Then HeraBEAT™ Intervention Group | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 24 | 52
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (4.5) | 30.0 (3.3) | 30.1 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 24 | 52
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 27 | 24 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 25 | 23 | 48
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Device Ease of Use
Description: Measured using the self-reported System Usability Scale (SUS) on 10 items, each on a scale from 1 to 5 (1 = strongly disagree and 5= strongly agree). A composite score is calculated with a range of 0-100 where higher values indicated a high usability of device, whereas lower scores indicate less usability of the device.
Time Frame: 8 weeks
Population: As this is a crossover trial, all patients participate in both arms. The arms above indicate the first intervention they are randomized to. The survey was administered after completion of each intervention group, this is why the number of participants is larger.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HeraBEAT™ Intervention Group | Standard Fetal Doppler Group
Number analyzed (Participants) | 52 | 51
score on a scale | 72.8 (19.1) | 75.1 (22.5)
Statistical Analysis 1: Comparison: HeraBEAT™ Intervention Group vs Standard Fetal Doppler Group; Difference in ease of use between our standard fetal Doppler and HeraBEAT™ device, as measured by the System Usability Survey (SUS) will be the primary outcome. We aim to recruit 50 participants (50 per arm, with cross-over) for a 99.7% power to detect a 10-point difference in SUS, as this accounts for a withdraw / post-randomization exclusion as high as 10% (assuming a proportion of expectant mothers to withdraw participation after being enrolled or found to not meet criteria after the fact); Test type: Superiority; p = 0.64, Regression, Linear; A generalized linear model adjusting by intervention group and the order of randomization was conducted; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-10.2 to 6.1]

2. Primary Outcome: Accurate Fetal Heart Rate Detection Where Values Are Between 110 and 160 Bpm
Description: Number of patients to detect a fetal heart rate accurately using the device. An inaccurate assessment is considered any value less than 110 or greater than 160 bpm. A patient with at least one inaccurate value is counted as an event of interest. Patients without an inaccurate event will be counted as a success.
Time Frame: 8 weeks
Population: As this study is a crossover study, all patients participate in each intervention group. The number analyzed reflects the number of participants that had fetal heart rate detection when they were participating in that group.
Measure: Count of Participants; unit: Participants
Arm/Group | HeraBEAT™ Intervention Group | Standard Fetal Doppler Group
Number analyzed (Participants) | 52 | 52
Participants | 40 | 42
Statistical Analysis 1: Comparison: HeraBEAT™ Intervention Group vs Standard Fetal Doppler Group; Test type: Superiority; p = 0.63, Chi-squared; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.57 to 2.53]

ADVERSE EVENTS:
Time Frame: Up to 37 weeks, which includes 6-8 weeks postpartum.
Description: For the crossover study, adverse events were monitored during the initial group the patient was assigned to as well as the intervention they crossed over to. Therefore, all patients enrolled are evaluated for adverse events in both intervention groups.
Arm/Group | HeraBEAT™ Intervention Group | Standard Fetal Doppler Group
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 0/52 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT04232215/Prot_SAP_000.pdf